CLINICAL TRIAL: NCT02706158
Title: Testing the Effect of a Dietary Intervention Program on the Incidence of Pre-eclampsia in Women at Risk
Brief Title: Dietary Intervention Program for Pre-eclampsia in Women at Risk
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Rambam Health Care Campus (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 310-15
Record Dates: First submitted 2016-02-28; First posted 2016-03-11 (Estimated); Last update posted 2016-03-15 (Estimated); Status verified 2016-03

CONDITIONS: Pre-eclampsia
MeSH Terms: conditions — Pre-Eclampsia | interventions — Calcium; Vitamin D; Dietary Supplements; Diet; Pregnancy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- supplement and balanced diet (Experimental): Woman at high risk of pre-eclampsia:
  supplements. 1500 mg Calcium and 1200 IU Vitamin D for 2 months. balanced diet.
  Interventions: Dietary Supplement: 1500 mg Calcium and 1200 IU Vitamin D for 2 months; Behavioral: balanced diet
- women without nutrition or supplement intervention (No Intervention): usual follow-up in the gynecology out patient clinic, without nutrition or supplement intervention.

INTERVENTIONS:
Dietary Supplement: 1500 mg Calcium and 1200 IU Vitamin D for 2 months — 1500 mg Calcium and 1200 IU Vitamin D for 2 months
  Other Names: supplement
  Arms: supplement and balanced diet
Behavioral: balanced diet — participants will get a balanced diet according to pregnancy stage
  Other Names: diet for pregnancy
  Arms: supplement and balanced diet

SUMMARY:
Aims: Pre-eclampsia is one of the leading causes of maternal and perinatal morbidity and mortality worldwide. Preeclampsia frequency is 2-8% from all pregnancies. Dietary factors and dietary status have been suggested to play a role in development of preeclampsia. Low intake of nutrients such as calcium, vitamin D, magnesium, omega 3 fatty acids, is related to increased risk of preeclampsia. Also high triglyceride levels, high BMI, low Omega 6: omega 3 ratio and high calories consumption are possible risk factors.

Material and Methods: A prospective study will be carried out. Woman medically diagnosed as high risk for preeclampsia will randomly be assigned to dietary treatment or no dietary treatment groups. In the dietary treatment group, besides medical care, all woman will get calcium and vitamin D supplementation from 8th to 16th gestational weeks, and thereafter until delivery personal extensive nutritional guidance. A 3 day food diary will be collected at inclusion and thereafter at Gestational weeks 16 and 28. All routinely collected data during pregnancy (blood tests, weight, blood pressure and preeclampsia symptoms) will be documented.

In both groups incidence of pre-eclampsia and eclampsia, blood pressure and protein in urine will be recorded.

DETAILED DESCRIPTION:
Aims: Pre-eclampsia is one of the leading causes of maternal and perinatal morbidity and mortality worldwide. Preeclampsia frequency is 2-8% from all pregnancies. Dietary factors and dietary status have been suggested to play a role in development of preeclampsia. Low intake of nutrients such as calcium, vitamin D, magnesium, omega 3 fatty acids, is related to increased risk of preeclampsia. Also high triglyceride levels, high BMI, low Omega 6: omega 3 ratio and high calories consumption are possible risk factors.

Material and Methods: A prospective study will be carried out. Woman medically diagnosed as high risk for preeclampsia will randomly be assigned to dietary treatment or no dietary treatment groups. In the dietary treatment group, besides medical care, all woman will get calcium and vitamin D supplementation from 8th to 16th gestational weeks, and thereafter until delivery personal extensive nutritional guidance. A 3 day food diary will be collected at inclusion and thereafter at Gestational weeks 16 and 28. All routinely collected data during pregnancy (blood tests, weight, blood pressure and preeclampsia symptoms) will be documented.

In both groups incidence of pre-eclampsia and eclampsia, blood pressure and protein in urine will be recorded.

ELIGIBILITY:
Inclusion Criteria:

* high risk of preeclampsia

Exclusion Criteria:

* age below 18
* low risk of preeclampsia

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 120 (Estimated)
Dates: Start 2016-04; Primary Completion 2017-04 (Estimated); Study Completion 2018-04 (Estimated)

PRIMARY OUTCOMES:
lower incidence of pre-eclampsia during pregnancy | up to 42 weeks gestation
lower incidence of pre-eclampsia post-partum | 4 weeks post delivery

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wang A, Rana S, Karumanchi SA. Preeclampsia: the role of angiogenic factors in its pathogenesis. Physiology (Bethesda). 2009 Jun;24:147-58. doi: 10.1152/physiol.00043.2008. PMID 19509125
- [Background] Duckitt K, Harrington D. Risk factors for pre-eclampsia at antenatal booking: systematic review of controlled studies. BMJ. 2005 Mar 12;330(7491):565. doi: 10.1136/bmj.38380.674340.E0. Epub 2005 Mar 2. PMID 15743856
- [Background] Oken E, Ning Y, Rifas-Shiman SL, Rich-Edwards JW, Olsen SF, Gillman MW. Diet during pregnancy and risk of preeclampsia or gestational hypertension. Ann Epidemiol. 2007 Sep;17(9):663-8. doi: 10.1016/j.annepidem.2007.03.003. Epub 2007 May 23. PMID 17521921
- [Background] Wei SQ, Audibert F, Hidiroglou N, Sarafin K, Julien P, Wu Y, Luo ZC, Fraser WD. Longitudinal vitamin D status in pregnancy and the risk of pre-eclampsia. BJOG. 2012 Jun;119(7):832-9. doi: 10.1111/j.1471-0528.2012.03307.x. Epub 2012 Mar 29. PMID 22462640
- [Background] Mehendale S, Kilari A, Dangat K, Taralekar V, Mahadik S, Joshi S. Fatty acids, antioxidants, and oxidative stress in pre-eclampsia. Int J Gynaecol Obstet. 2008 Mar;100(3):234-8. doi: 10.1016/j.ijgo.2007.08.011. Epub 2007 Oct 31. PMID 17977540
- [Background] Clausen T, Slott M, Solvoll K, Drevon CA, Vollset SE, Henriksen T. High intake of energy, sucrose, and polyunsaturated fatty acids is associated with increased risk of preeclampsia. Am J Obstet Gynecol. 2001 Aug;185(2):451-8. doi: 10.1067/mob.2001.116687. PMID 11518908
- [Background] Kanagal DV, Rajesh A, Rao K, Devi UH, Shetty H, Kumari S, Shetty PK. Levels of Serum Calcium and Magnesium in Pre-eclamptic and Normal Pregnancy: A Study from Coastal India. J Clin Diagn Res. 2014 Jul;8(7):OC01-4. doi: 10.7860/JCDR/2014/8872.4537. Epub 2014 Jul 20. PMID 25177604